CLINICAL TRIAL: NCT02070575
Title: Evaluation of Molecular Forms of PSA and Human Kallikrein 2 in a Cohort of Patients With Locally Resected Prostate Cancer But Biochemical Recurrence
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 14-041
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Prostate Cancer
Keywords: PSA; Human Kallikrein 2; locally resected prostate cancer; biochemical recurrence; 14-041
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Blood sample

GROUPS / COHORTS (1):
- Pts with prostate cancer: This study is planned to determine the kallikrein panel of 200 patients presenting with biochemical recurrence (PSA ≥ 0.05ng/ml) after radical prostatectomy prior to any additional therapy or minimum post 1 year additional therapy.
  Interventions: Other: blood draw

INTERVENTIONS:
Other: blood draw — Venous blood will be collected in an EDTA Vacutainer tubeup to 10 mL and will be immediately put on ice. This sample may be drawn as a stand-alone blood draw. Samples will be centrifuged at 1900g (3000-3200 RPM) for 15 Minutes and the serum aliquoted into freezer vials and stored at -80°C until analysis. In addition patients who have not received treatment for biochemical recurrence after their first draw are eligible for subsequent draws to determine the reproducibility of the test over time.

SUMMARY:
The purpose of this study is to investigate if a new blood test looking at PSA and a group of PSA related proteins in a patient's blood can indicate which men after surgery with a rising PSA could benefit from treatment, and/or indicate which men are at higher risk for recurrence before initial treatment is given.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with radical prostatectomy that develop a rising serum PSA ≥ 0.05ng/ml and have not received any kind of additional therapy.
* Patients who have had additional therapy post radical prostatectomy are eligible for this study if ≥1 year has passed since treatment and the patient develops a rising serum PSA ≥0.05ng/ml.

Exclusion Criteria:

* Previous additional therapy for prostate cancer, less than 1 year ago
* No evidence of rising PSA
* Patients unwilling to undergo venesection

Min Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment, the protocol investigator, or research team at Memorial Sloan Kettering Cancer Center (MSKCC).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-02-20 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
profile of a panel of kallikrein related serine proteases in the blood | 2 years
  of patients that present with biochemical recurrence after radical prostatectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Laudone, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/